CLINICAL TRIAL: NCT07176741
Title: Measurement of Hepatocyte TREM-1 Expression Level to Evaluate Its Intrinsic Performance and Prognostic Value in Severe Symptomatic Alcohol-related Hepatitis
Brief Title: LiverTREM-1: Hepatic TREM-1 Expression and Prognosis in Severe Alcoholic Hepatitis
Acronym: Liver TREM-1
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, HAGHNEJAD Vincent, Dr, Central Hospital, Nancy, France
Other Study IDs: 2023PI101
Record Dates: First submitted 2025-06-15; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Severe Alcoholic Hepatitis
Keywords: TREM-1; sAH; biomarker; prognosis; alcoholic hepatitis; alcohol use disorder; AUD; cirrhosis
MeSH Terms: conditions — Hepatitis, Alcoholic; Alcoholism; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — histological staining
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biopsy-proven severe alcoholic hepatitis and control liver specimens: Cases: Adults treated at CHRU de Nancy (2013-2023) for Severe Alcoholic Hepatitis, with archived liver biopsies.
  Controls: Adults with liver malignancies and archived biopsies.
  Interventions: Diagnostic Test: TREM-1 expression (via immunohistochemistry) between SAH patients and controls

INTERVENTIONS:
Diagnostic Test: TREM-1 expression (via immunohistochemistry) between SAH patients and controls — this is the first study to focus on hepatocyte-specific TREM-1 expression in human liver tissue
  What Distinguishes This Study Tissue-Level Focus: Unlike most studies that assess blood biomarkers or systemic inflammation, this research directly measures TREM-1 expression in liver tissue (hepatocytes), offering localized insights into disease severity and immune response.
  Retrospective Biobank Utilization: Leverages a rich biobank of archival biopsies spanning 10 years, ensuring real-world data and long-term clinical follow-up-rarely combined at this scale in similar research.
  Dual Purpose (Diagnostic & Prognostic): Most biomarkers are evaluated for either diagnostic or prognostic value-this study uniquely addresses both in a single, comprehensive framework.
  Therapeutic Translation Potential: TREM-1 is already a target for pharmacological inhibition (e.g., with peptide inhibitors tested safely in humans for other conditions). This positions the study for rapid clinical translation,

SUMMARY:
Background & Rationale Severe alcohol-related hepatitis (SAH) is a serious condition with a 3-month mortality rate of ~30%. Diagnosis and prognosis are complex due to non-specific and insensitive clinical, biological, and histological indicators. Corticosteroids-the only validated treatment-are only effective in 50% of cases and can worsen outcomes in non-responders by promoting infections. Liver transplantation remains a limited option due to organ scarcity and patient eligibility.

TREM-1, a pro-inflammatory receptor, has shown promise in inflammatory liver diseases. Its expression in hepatocytes may serve as a biomarker to better classify patients, guide treatment, and improve outcomes.

Objectives

Primary Objective:

Compare TREM-1 expression (via immunohistochemistry) between SAH patients and controls with other liver diseases (e.g., HCC, metastatic colon cancer, cholangiocarcinoma).

Secondary Objectives:

Determine optimal antibody dilution for TREM-1 staining.

Assess diagnostic performance (sensitivity, specificity, PPV, NPV).

Identify homogeneous SAH subgroups using clinical, histological, and biological data.

Evaluate prognostic value of TREM-1 expression for:

2-month mortality

Corticosteroid response (bilirubin regression at Day 7)

Lille score <0.45 at Day 7

Compare TREM-1's predictive power to standard scores (MELD, Maddrey, Lille, etc.).

Methodology

Population:

Cases: Adults treated at CHRU de Nancy (2013-2023) for SAH, with archived liver biopsies.

Controls: Adults with liver malignancies and archived biopsies.

Sample Size:

Phase I: 12 cases, 6 controls

Phase II: 150 cases, 150 controls

Data Sources: Medical records, archived pathology slides

Statistical Tools: Logistic regression, survival analysis, ROC curves, clustering, SAS/R software

Expected Outcomes & Impact Improved prognostic stratification and therapeutic guidance for SAH patients

Better targeting of corticosteroid therapy to reduce unnecessary risk

Early referral for liver transplantation when appropriate

Validation of TREM-1 as a diagnostic/prognostic biomarker

Foundation for future TREM-1-targeted clinical trials

Potential paradigm shift linking liver histology with real-time clinical decision-making

Enhanced resource allocation and patient management

DETAILED DESCRIPTION:
Study Title

Official Title:

Liver TREM-1: Hepatic Expression of TREM-1 in Severe Alcoholic Hepatitis

Brief Summary (250 words max) Severe alcohol-associated hepatitis (sAH) is a life-threatening liver disease with a 3-month mortality rate of up to 30%. The only validated treatment-corticosteroids-fails in approximately 40% of patients, increases infection risk, and offers no survival benefit beyond 28 days. Therefore, there is an urgent need to identify prognostic biomarkers to guide therapy.

TREM-1 (Triggering Receptor Expressed on Myeloid cells 1) is a pro-inflammatory receptor expressed on hepatic immune and endothelial cells. Preclinical murine studies suggest it plays a pivotal role in alcohol-induced liver injury. This observational study aims to assess the diagnostic and prognostic value of hepatic TREM-1 expression in patients with severe alcohol-associated hepatitis using archived liver biopsy samples.

A total of 300 archived liver specimens (150 sAH cases, 150 controls with hepatic malignancies) will be analyzed via immunohistochemistry using a validated TREM-1 scoring system. Outcomes include TREM-1 expression levels, correlation with clinical parameters, mortality at 2 months, and response to corticosteroid therapy.

Detailed Description The study will determine whether hepatic TREM-1 expression can serve as a biomarker to stratify sAH patients into prognostic subgroups. TREM-1 expression will be measured via immunostaining and categorized as high vs. low using a score developed by Duan et al. Secondary analyses include diagnostic accuracy, treatment response (based on jaundice regression and Lille score at Day 7), and survival at 2 months. Statistical models (logistic regression, survival analysis, ROC curves, clustering) will be used.

This study complies with the Declaration of Helsinki, EU Regulation 536/2014, MR004 guidelines (CNIL), and French Public Health laws 2004-806, 2004-800, and 2016-41.

Study Type Observational

Observational Model: Cross-sectional

Time Perspective: Retrospective

Biospecimen Retention: Samples retained (Slides; No DNA)

Primary Outcome Measure Hepatic TREM-1 Expression

Type: Binary categorical variable (high vs. low)

Time Frame: At the day of liver biopsy

Method: Immunohistochemistry (Duan et al. score)

Secondary Outcome Measures Diagnostic Accuracy of TREM-1

Sensitivity, specificity, PPV, NPV for sAH diagnosis

Gold standard: multidisciplinary diagnosis

Time Frame: at the day of liver biopsy

Jaundice Resolution

Binary variable: resolved/persistent at Day 7

Time Frame: 7 days after corticosteroid start

Lille Score < 0.45

Prognostic response to corticosteroids

Time Frame: Day 7

Mortality at 2 Months

Time Frame: 60 days post-diagnosis

Analysis: Cox regression

Cluster Analysis of sAH Subgroups

Based on TREM-1 expression and clinico-biological profiles

Comparison to Established Prognostic Scores

MELD, AHHS, Glasgow, Maddrey, SALVE, Lille, Lille-MELD

TREM-1 expression in RNAseq3' in SAH patients

categorical variable (detected vs undetected) and quantitative variable (TREM expression as fragments per millions)

Comparison of TREM-1 expression in RNAseq3' in SAH patients to prognostic scores and outcomes

MELD, AHHS, Glasgow, Maddrey, SALVE, Lille, Lille-MELD Infection from day 3 to day 180 Mortality at M2, M3 and M6 Overall Mortality Response to steroids

Enrollment Estimated Enrollment: 300

Sampling Method: Non-probability sample

Eligibility Criteria

Inclusion Criteria (Cases):

Adults (≥18) with biopsy-proven severe alcohol-associated hepatitis (2013-2024)

Available liver biopsy slides at CHRU Nancy

Non-opposition documented

Inclusion Criteria (Controls):

Adults (≥18) with hepatic resection for colorectal metastases, cholangiocarcinoma, or HCC

Archived liver samples available

Non-opposition documented

Exclusion Criteria:

No histologic diagnosis of sAH

Depleted paraffin blocks unsuitable for staining

Study Dates Start Date: Upon ethics approval

Primary Completion Date: ~9 months after start

Study Completion Date: ~15 months after start

Locations CHRU Nancy, France Lead Pathology and Hepatology Units Collaborating Site: Hôpital Henri Mondor (AP-HP)

Sponsor and Contacts Sponsor: CHRU Nancy Scientific PI: Dr. Vincent Haghnejad Email: v.haghnejad@chru-nancy.fr Phone: +33 625150180

Regulatory Compliance

This study adheres to the following regulations and ethical standards:

Declaration of Helsinki

EU Regulation (EU) 536/2014

French Public Health Law: 2004-806, 2004-800, 2016-41

Bioethics Law and GDPR (EU 2016/679)

CNIL MR004 framework for retrospective, non-interventional data use

Statistical Methods

Primary Objective:

Logistic regression (univariate p<0.2 threshold, stepwise multivariate model) to compare TREM-1 expression between cases and controls.

Secondary Objectives:

ROC curve analysis to determine optimal antibody dilution (AUC, Youden index).

Diagnostic accuracy metrics (sensitivity, specificity, PPV, NPV).

Clustering (Multiple Correspondence Analysis + Ward's Hierarchical Clustering) for subgroup discovery.

Cox model for 2-month mortality.

Logistic regression for treatment response (Day 7 jaundice, Lille score <0.45).

Comparative model performance vs. MELD, Maddrey, etc.

Software: SAS 9.4 or R

Significance Level: 5% (two-sided)

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Individuals who received full information about the study and did not object to the use of their data within this research.
* Patients managed in one of the intensive care or hepatogastroenterology departments at CHRU de Nancy for severe alcohol-related hepatitis between January 1, 2013, and December 31, 2023.
* Archived liver biopsy slides available at CHRU de Nancy.
* Adult patients at the time of diagnosis.

Controls:

* Individuals who received full information about the study and did not object to the use of their data within this research.
* Patients treated and operated on at CHRU de Nancy for hepatocellular carcinoma, colorectal cancer liver metastasis, or cholangiocarcinoma between January 1, 2013, and December 31, 2023.
* Archived liver biopsy slides available at CHRU de Nancy.
* Adult patients at the time of diagnosis.

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case:
  Adult patient managed in one of the intensive care or hepatogastroenterology departments at CHRU de Nancy for severe alcohol-related hepatitis between January 1, 2013, and December 31, 2023, inclusive.
  Control:
  Adult patient managed and operated on at CHRU de Nancy for hepatocellular carcinoma, colorectal cancer liver metastasis, or cholangiocarcinoma between January 1, 2013, and December 31, 2023, inclusive.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Hepatocyte TREM-1 expression in SAH patients vs. controls on the day of biopsy | Day 0 index liver biopsy
  Compare hepatocyte TREM-1 expression (via immunohistochemistry) in patients with severe alcohol-associated hepatitis (SAH) versus controls with other liver diseases (e.g., hepatocellular carcinoma, colorectal liver metastases, cholangiocarcinoma). TREM-1 expression is scored as high or low using a validated semi-quantitative method.
  Unit of Measure: Median hepatocyte TREM-1 H-score [IQR] Archival liver specimens obtained Jan 1, 2013-Dec 31, 2024 were used; assessment reflects baseline (the day of the biopsy).

SECONDARY OUTCOMES:
Baseline TREM-1 expression (via RNAseq3') in patients with severe alcohol-associated hepatitis (SAH) | Day 0 (index liver biopsy)
  Compare hepatocyte TREM-1 expression (via RNAseq3') in patients with severe alcohol-associated hepatitis (SAH). TREM expression is normalized according to sequencing depth and gene length.
  Median hepatocyte TREM-1 [IQR] or mean +/- [SD] and Binary detection of hepatocyte TREM-1 by 3' RNA-seq. Expressor (Detected) = normalized transcript value > 0 (e.g., FPM > 0); Non-expressor (Not detected) = 0.
  RNA was extracted from tissue taken at the baseline biopsy; archival specimens span Jan 1, 2013-Dec 31, 2024.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Haghnejad, MD, Principal Investigator — CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duan M, Wang ZC, Wang XY, Shi JY, Yang LX, Ding ZB, Gao Q, Zhou J, Fan J. TREM-1, an inflammatory modulator, is expressed in hepatocellular carcinoma cells and significantly promotes tumor progression. Ann Surg Oncol. 2015 Sep;22(9):3121-9. doi: 10.1245/s10434-014-4191-7. Epub 2014 Dec 3. PMID 25465376
- [Background] Ichou L, Carbonell N, Rautou PE, Laurans L, Bourcier S, Pichereau C, Baudel JL, Nousbaum JB, Renou C, Anty R, Tankovic J, Maury E, Guidet B, Landraud L, Ait-Oufella H. Ascitic fluid TREM-1 for the diagnosis of spontaneous bacterial peritonitis. Gut. 2016 Mar;65(3):536-8. doi: 10.1136/gutjnl-2015-310160. Epub 2015 Jul 3. No abstract available. PMID 26141143
- [Background] Francois B, Lambden S, Garaud JJ, Derive M, Grouin JM, Asfar P, Darreau C, Mira JP, Quenot JP, Lemarie J, Mercier E, Lacherade JC, Vinsonneau C, Fivez T, Helms J, Badie J, Levy M, Cuvier V, Salcedo-Magguilli M, Laszlo-Pouvreau AL, Laterre PF, Gibot S; ESSENTIAL investigators. Evaluation of the efficacy and safety of TREM-1 inhibition with nangibotide in patients with COVID-19 receiving respiratory support: the ESSENTIAL randomised, double-blind trial. EClinicalMedicine. 2023 Jun;60:102013. doi: 10.1016/j.eclinm.2023.102013. Epub 2023 May 31. PMID 37350989
- [Background] Francois B, Lambden S, Fivez T, Gibot S, Derive M, Grouin JM, Salcedo-Magguilli M, Lemarie J, De Schryver N, Jalkanen V, Hicheur T, Garaud JJ, Cuvier V, Ferrer R, Bestle M, Pettila V, Mira JP, Bouisse C, Mercier E, Vermassen J, Huberlant V, Vinatier I, Anguel N, Levy M, Laterre PF; ASTONISH investigators. Prospective evaluation of the efficacy, safety, and optimal biomarker enrichment strategy for nangibotide, a TREM-1 inhibitor, in patients with septic shock (ASTONISH): a double-blind, randomised, controlled, phase 2b trial. Lancet Respir Med. 2023 Oct;11(10):894-904. doi: 10.1016/S2213-2600(23)00158-3. Epub 2023 May 31. PMID 37269870
- [Background] Francois B, Wittebole X, Ferrer R, Mira JP, Dugernier T, Gibot S, Derive M, Olivier A, Cuvier V, Witte S, Pickkers P, Vandenhende F, Garaud JJ, Sanchez M, Salcedo-Magguilli M, Laterre PF. Nangibotide in patients with septic shock: a Phase 2a randomized controlled clinical trial. Intensive Care Med. 2020 Jul;46(7):1425-1437. doi: 10.1007/s00134-020-06109-z. Epub 2020 May 28. PMID 32468087
- [Background] Mathurin P, Duchatelle V, Ramond MJ, Degott C, Bedossa P, Erlinger S, Benhamou JP, Chaput JC, Rueff B, Poynard T. Survival and prognostic factors in patients with severe alcoholic hepatitis treated with prednisolone. Gastroenterology. 1996 Jun;110(6):1847-53. doi: 10.1053/gast.1996.v110.pm8964410.